CLINICAL TRIAL: NCT05007353
Title: The SINgapore GERiatric Intervention Study to Reduce Cognitive Decline and Physical Frailty (SINGER) Study, Biomarker and Health Service Research Analyses
Brief Title: The SINgapore GERiatric Intervention Study to Reduce Cognitive Decline and Physical Frailty (SINGER) Study
Acronym: SINGER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University of Singapore (Other)
Collaborators: National Medical Research Council (NMRC), Singapore (Other Government)
Responsible Party: Principal Investigator, Christopher Chen Li-Hsian, Associate Professor, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SINGER 2021
Record Dates: First submitted 2021-07-28; First posted 2021-08-16 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Cognitive Impairment; Alzheimer Disease; Vascular Cognitive Impairment; Dementia; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Neurocognitive Disorders; Mental Disorders; Cognition Disorder
Keywords: cognitive decline; cognitive impairment; multi-domain lifestyle interventions; dementia; elderly
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease; Dementia; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Neurocognitive Disorders; Mental Disorders; Cognition Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Structured Lifestyle Intervention (Experimental): Structured lifestyle modification program developed for participants targeting diet, physical exercise, cognitive training, and social stimulation.
  Interventions: Behavioral: Structured Lifestyle Intervention
- Self-Guided Intervention (Experimental): General health information provided to participants.
  Interventions: Behavioral: Self-Guided Intervention

INTERVENTIONS:
Behavioral: Structured Lifestyle Intervention — Structured Lifestyle Intervention (SLI) involves providing participants with intensive structure and support by a team of trainers to increase physical exercise, adhere to a healthy diet, cognitive training, increase intellectual/social stimulation, and better manage vascular risk factors.
  Other Names: SLI
  Arms: Structured Lifestyle Intervention
Behavioral: Self-Guided Intervention — In the Self-Guided Intervention (SGI), education about the importance of a healthy lifestyle as a preventive strategy and support to encourage change will be provided.
  Other Names: SGI
  Arms: Self-Guided Intervention

SUMMARY:
A study in Finland found that a multidomain intervention of physical activity, nutritional guidance, cognitive training, social activities and management of vascular risk factors slowed cognitive decline in healthy older adults at increased risk of cognitive decline. A 6-month pilot study was initiated in Singapore, which demonstrated the cultural feasibility and practicality of the FINGER interventions and a set of locally adapted interventions in an Asian population. The SINGER study is a 2-year randomized controlled trial that aims to test the efficacy and safety of these lifestyle changes, including diet and cardiovascular risk factor management, cognitive and physical exercises, in delaying cognitive decline in older adults at risk of dementia.

DETAILED DESCRIPTION:
Results from a population-based 2-year clinical trial, the Finnish Geriatric Intervention Study to Prevent Cognitive Impairment and Disability (FINGER), demonstrated that a multidomain intervention of physical activity, nutritional guidance, cognitive training, social activities and management of vascular risk factors slowed cognitive decline in healthy older adults at increased risk of cognitive decline. Currently, no pharmacological treatment options that can rival these effects. Thus, there is an urgent need to test the generalizability, adaptability, and sustainability of these findings in Singaporean populations. A 6-month pilot study was initiated in Singapore, which demonstrated the cultural feasibility and practicality of the FINGER interventions and a set of locally adapted interventions in an Asian population. Hence, the next step was to conduct a larger scale SINGER trial to determine the efficacy of these interventions in Singapore. If the interventions are found to be effective and safe with high applicability and scalability, the study will provide important clinical and public health implications to a rapidly increasing ageing population.

ELIGIBILITY:
Inclusion Criteria:

* Age 60-77 years
* Able to understand English/Chinese
* Risk of dementia: Cardiovascular Risk Factors, Aging, and Incidence of Dementia (CAIDE) dementia risk score >6 indicating the presence of modifiable risk factors Modifiable lifestyle factors (fulfilling at least one of the following LIBRA index for diet, cognitive activity, physical activity)
* Cognitive performance at the mean level or slightly lower than expected for age (MoCA ≥18, ≤27)
* No plans to travel outside of Singapore for an extended period of time over the course of the study
* Free of physical disabilities that preclude participation in the study
* Willing to complete all study-related activities for 24 months
* Willing to be randomized to either lifestyle intervention group

Exclusion Criteria:

* malignant diseases
* dementia
* substantial cognitive decline (MoCA<18)
* major depression
* symptomatic cardiovascular disease
* revascularisation within 1 year
* severe loss of vision, hearing or communicative ability
* other conditions inhibiting from safe engagement in the prescribed intervention and other conditions preventing cooperation, as judged by the study physician

Ages: 60 Years to 77 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2021-08-23 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Global Cognition | Up to 2 years
  Global cognition measured using the modified Neuropsychological Test Battery (mNTB) that includes: Visual Paired Associates, Logical Memory Recall of the Wechsler Memory Scale-Revised, Rey Auditory Verbal Learning, Digit Span, Word and Category Fluency test, Trail Making Test, Letter Digit Substitution test.

SECONDARY OUTCOMES:
Episodic Memory | Up to 2 years
  Episodic memory measured using mNTB subtests: Visual paired associates tests, Logical Memory immediate and delayed recall of the Wechsler Memory Scale-Revised, Rey Auditory Verbal Learning test.
Executive Function | Up to 2 years
  Executive function measured using mNTB subtests: Digit Span, Word and Category Fluency test, Trail Making Test Part B.
Processing Speed | Up to 2 years
  Processing speed measured using mNTB subtests: Letter Digit Substitution test and Trail-Making Test Part A.
Clinical Dementia Rating-Sum of Boxes (CDR-SB) | Up to 2 years
  The Clinical Dementia Rating-Sum of Boxes (CDR-SB) is scored from 0 to 18. Higher scores reflect worse performance.
Alzheimer's Disease Cooperative Study Activities of Daily Living-Mild Cognitive Impairment-Activities of Daily Living Inventory (ADCS-MCI-ADL) | Up to 2 years
  The Alzheimer's Disease Cooperative Study Activities of Daily Living-Mild Cognitive Impairment-Activities of Daily Living Inventory (ADCS-MCI-ADL) is scored from 0 to 53. Higher scores reflect better performance.
The Geriatric Depression Scale (GDS) | Up to 2 years
  The Geriatric Depression Scale (GDS) is scored from 0 to 15. Scores of 0-4 are considered normal, 5-8 indicate mild depression; 9-11 indicate moderate depression; and 12-15 indicate severe depression.
Global Physical Activity Questionnaire (GPAQ) | Up to 2 years
  The Global Physical Activity Questionnaire (GPAQ) measures physical activity across 3 domains: work, travel, and recreation, as well as average time per day spent in sedentary behavior. The GPAQ is scored based on a population's mean or median physical activity spent in physical activity or by classifying a certain percentage of a population as 'inactive' or 'insufficiently active'.
Prospective-Retrospective Memory Questionnaire | Up to 2 years
  The Prospective-Retrospective Memory Questionnaire (PRMQ) is measured on a 5-point scale. Higher scores represent greater frequency of memory failures.
Pittsburgh Sleep Quality Index (PSQI) | Up to 2 years
  The Pittsburgh Sleep Quality Index (PSQI) is scored from 0 to 21. Higher scores indicate worse sleep quality.
Leisure-Time Activities Questionnaire | Up to 2 years
  The Leisure-Time Activities Questionnaire measures the frequency of engagement in the following activities: Health activities, Social activities, Productive activities, Fitness activities, Recreational activities, Any cognitively-stimulating activities. Scores are measured on a 3-point scale. Higher scores represent higher frequency of engagement in leisure-time activities.
Physical Performance Test (PPT) | Up to 2 years
  The Physical Performance Test (PPT) is scored from 0 to 36. Higher scores represent better performance.
Quality of Life Questionnaire (15D) | Up to 2 years
  The Quality of Life Questionnaire (15D) has a single index (15D score) on a 0-1 scale, which represents overall HRQoL (0 = being dead, 0.0162 = being unconscious or comatose, 1 = no problems on any dimension = 'full' HRQOL). This is calculated from the health state descriptive system by using a set of population-based preference or utility weights.
36-Item Short Form Survey (SF-36) | Up to 2 years
  The 36-Item Short Form Survey (SF-36) has eight domains. Each domain is scored from 0 to 100. Higher scores represent a more favourable health state.
Resource Use Inventory (RUI) | Up to 2 years
  The Resource Use Inventory (RUI) measures 4 domains: direct medical care, direct nonmedical care, informal care, and subjects' time use. The RUI is filled in based on the frequency and amount of resources used. If none were used, '00' is entered.
Height | Up to 2 years
  Height is measured in metres.
Weight | Up to 2 years
  Weight is measured in kilograms.
Hip and waist circumference | Up to 2 years
  Hip and waist circumference measured in centimetres.
Changes in Blood Pressure | Up to 2 years
  Vascular and metabolic risk factors measured by changes in blood pressure in mmHg. Incident events using serious adverse event reports will also be assessed.
Changes in Lipid Profile | Up to 2 years
  Vascular and metabolic risk factors measured by changes in lipid profile in mmol/L.
Changes in Glucose Regulation | Up to 2 years
  Vascular and metabolic risk factors measured by changes in glucose regulation in mmol/L.
Neuroimaging | Up to 2 years
  Magnetic Resonance Imaging will be used to assess changes in brain structural integrity, grey matter volume loss, white matter microstructure degradation, and increase of cerebrovascular disease markers (CeVD). Vascular polygenic risk scores (PRS) and its association with neurodegeneration, CeVD burden and cognitive decline will be performed.
Blood Biomarkers | Up to 2 years
  Novel and accessible blood markers to monitor AD- and CeVD-associated pathologies will be measured. Plasma concentrations of cardiac markers (High-sensitive cardiac troponin T (hs Troponin T), N-terminal pro b-type natriuretic peptide (NT-proBNP) and Growth/differentiation factor 15 (GDF 15)), and peripheral biomarkers of Aβ, tau and synaptic pathology, oxidative stress, endothelial/cardiovascular injury and degenerative protein modifications (DPMs) damaged proteins will be used.
Retinal Imaging Markers | Baseline only
  Multimodal retinal imaging will be used to assess retinal structural, vascular and neuronal changes.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher LH Chen, MD, Principal Investigator — National University of Singapore
Locations (3):
- Singapore (3):
  - National University Hospital, Singapore
  - National University of Singapore, Yong Loo Lin School of Medicine, Singapore
  - National Neuroscience Institute @ Tan Tock Seng Campus (NNI @ TTSH campus), Singapore

IPD SHARING:
Plan to Share IPD: No
Interested collaborators may put in a request.

REFERENCES:
- [Background] Ngandu T, Lehtisalo J, Solomon A, Levalahti E, Ahtiluoto S, Antikainen R, Backman L, Hanninen T, Jula A, Laatikainen T, Lindstrom J, Mangialasche F, Paajanen T, Pajala S, Peltonen M, Rauramaa R, Stigsdotter-Neely A, Strandberg T, Tuomilehto J, Soininen H, Kivipelto M. A 2 year multidomain intervention of diet, exercise, cognitive training, and vascular risk monitoring versus control to prevent cognitive decline in at-risk elderly people (FINGER): a randomised controlled trial. Lancet. 2015 Jun 6;385(9984):2255-63. doi: 10.1016/S0140-6736(15)60461-5. Epub 2015 Mar 12. PMID 25771249
- [Background] Chew KA, Xu X, Siongco P, Villaraza S, Phua AKS, Wong ZX, Chung CY, Tang N, Chew E, Henry CJ, Koo E, Chen C. SINgapore GERiatric intervention study to reduce physical frailty and cognitive decline (SINGER)-pilot: A feasibility study. Alzheimers Dement (N Y). 2021 Mar 15;7(1):e12141. doi: 10.1002/trc2.12141. eCollection 2021. PMID 33748399